CLINICAL TRIAL: NCT04673578
Title: Celecoxib Versus Placebo as an Adjunct to Treatment-as-usual in Children and Youth With Obsessive-compulsive Disorder: A Single-site Randomized Quadruple-blind Phase II Study
Brief Title: Adjunctive Celecoxib in Childhood-onset OCD Study
Acronym: ACE-OCD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: BC Children's Hospital Research Institute (Other); Obsessive Compulsive Foundation (Other)
Responsible Party: Principal Investigator, Evelyn Stewart, MD, Professor, Division of Clinical & Behavioural Neurosciences, Department of Psychiatry, Faculty of Medicine; Medical Director, BCCH Provincial OCD Program (POP); Investigator, BC Children's Hospital, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H19-03886
Record Dates: First submitted 2020-11-24; First posted 2020-12-17 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Obsessive-Compulsive Disorder; Pediatric Psychiatric Disorder
Keywords: Non-steroidal anti-inflammatory drug; Cyclooxygenase inhibitor; Celecoxib; Inflammation; Children; Obsessive-compulsive disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Neurodevelopmental Disorders; Inflammation | interventions — Celecoxib

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to celecoxib or placebo arms. Participants will have the option of participating in a 12-week open-label celecoxib extension after completing the randomized portion of the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo capsules will be dispensed similar in appearance to celecoxib capsules. Unique randomization codes will be used for each participant to avoid inadvertent loss of blinding for all participants in the event that one is unblinded. Data analysis and manuscript writing will be performed after unblinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Celecoxib (Experimental): Celecoxib 50 mg orally twice daily (if weight 10-25 kg) or 100 mg orally twice daily (if weight > 25 kg) for 12 weeks. Used as adjunct to treatment-as-usual.
  Interventions: Drug: Celecoxib
- Placebo (microcrystalline cellulose) (Placebo Comparator): Placebo capsules identical to celecoxib. One capsule orally twice daily for 12 weeks. Used as adjunct to treatment-as-usual.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Celecoxib — Selective COX-2 inhibitor; nonsteroidal anti-inflammatory drug (NSAID)
  Other Names: MINT-CELECOXIB; NDC Code: 0025-1525; ATC Code: M01AH01; Canadian DIN: 02412497
  Arms: Celecoxib
Other: Placebo — Microcrystalline cellulose
  Arms: Placebo (microcrystalline cellulose)

SUMMARY:
This is a randomized, controlled, single-centre phase II superiority trial to determine the efficacy of 12 weeks of celecoxib (50 mg or 100 mg orally twice daily, dosed based on weight) compared to placebo as an adjunct to treatment-as-usual in children and youth with moderate-to-severe obsessive-compulsive disorder.

DETAILED DESCRIPTION:
Cyclooxygenase (COX) enzymes oxidize arachidonic acid to prostaglandins, which modulate normal neuronal function and inflammatory responses in the central nervous system. COX-2, which is constitutively expressed by glutamatergic neurons in the cortex, hippocampus, and amygdala, plays an important physiological role in synaptic plasticity and long-term potentiation. Pre-clinical studies point to a potential role for non-steroidal anti-inflammatory drugs (NSAIDs), which inhibit COX enzymes, in modulation of mood and anxiety symptoms. Recent meta-analyses also suggest a role for adjunctive COX inhibitors in the treatment of depression and first-episode schizophrenia. While consensus guidelines on the use of anti-inflammatory therapy in children with acute-onset subtypes of childhood-onset obsessive compulsive disorder (OCD) suggest NSAIDs as a first-line option for patients with mild impairment, there is limited empirical evidence to support their use in this population. Two small randomized-controlled trials in adults with OCD demonstrated improved symptom severity with celecoxib - a selective COX-2 inhibitor - raising the possibility that COX inhibition may be effective in a general OCD population.

The primary objective of this study is to compare the effects of celecoxib and placebo as adjuncts to treatment-as-usual on reduction in symptom severity, as determined by Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS) after 12 weeks in children and youth with moderate-to-severe OCD.

This is a randomized, controlled, single-centre superiority trial with two parallel groups (celecoxib 50 mg [≤25 kg] or 100 mg [>25 kg] twice daily and placebo). Participants will be recruited from the BC Children's Hospital (BCCH) Provincial OCD Program and based on self-referral from community practices. Randomization will be performed as block randomization with a 1:1 allocation and stratified based on pre-treatment symptom severity. The investigator, outcomes assessor, clinician, and patient will be blinded to the intervention groups. Labs at baseline and 12 weeks will include complete blood count (CBC) with differential, creatinine, electrolytes, liver enzymes, and CRP. Participants will be assessed for OCD severity and adverse events at weeks 6 and 12. Analysis will be carried out according to intention-to-treat principles. Power calculations using estimates based on previous studies suggest a target recruitment of 80 participants. Participants will be offered a 12-week open-label celecoxib extension following the blinded phase for further assessment of tolerability.

The primary outcome is OCD severity (as measured by total CY-BOCS score) after 12 weeks in the celecoxib compared to placebo arm, adjusted for baseline. Secondary outcomes include CY-BOCS score after 6 weeks adjusted for baseline OCD severity, difference in the proportion of participants achieving a clinically meaningful response or remission; mean clinical global impression of severity and improvement after 6 and 12 weeks; and difference between celecoxib and placebo arms in the proportion of participants reporting adverse events that are possibly, probably, or definitely related to the study intervention.

NSAIDs are common in clinical practice and referenced in both adult and pediatric treatment guidelines for OCD, but no controlled studies have evaluated the effects of COX inhibitors in childhood-onset OCD. This study will be the first to assess the efficacy and safety of adjunctive celecoxib in this population and will inform clinical management of children and youth with OCD.

ELIGIBILITY:
Inclusion Criteria:

1. Age 7-18 years
2. Resident of British Columbia
3. DSM-5 diagnosis of OCD based on (a) history of prior clinician assessment and (b) standardized interview
4. CY-BOCS score ≥16 (moderate to severe)
5. Able to take medication twice daily in capsule form (in whole form or sprinkled contents)
6. Negative pregnancy test (either serum or urine) in participants with child-bearing potential
7. Use of highly effective and/or double barrier contraception, or abstinence, in participants with child-bearing potential

Exclusion Criteria:

1. Lifetime diagnosis of renal disease, liver disease, gastrointestinal bleeding, peptic ulcer disease, inflammatory bowel disease, severe or uncontrolled asthma, bleeding disorders, heart disease, heart failure, or hypertension
2. Current major depressive episode, acute psychosis, active substance use, suicidality, or restriction of fluid intake
3. Pregnant or breastfeeding during the study period
4. Active infection or antibiotic treatment at baseline
5. Allergy to celecoxib, sulfonamide compounds, or NSAIDs, including aspirin
6. Current or previous regular use of immune-modulating therapies for treatment of OCD symptoms, at an effective anti-inflammatory dose (including NSAIDs, corticosteroids, or biologics)
7. Use of NSAIDs at any dose at a frequency ≥ 3 times per week during the 2 months prior to randomization
8. Current use of intravenous or oral corticosteroids
9. Concurrent use of CYP2C9 inhibitors fluconazole, amiodarone, oxandrolone or methotrexate; CYP2C9 inducers including rifampin and phenobarbital; or any other drug that may interact with celecoxib and, in the opinion of Dr. Stewart or another study investigator, represents a potential safety risk
10. Poor CYP2C9 metabolizer (i.e. CYP2C9*3/*3 genotype) based on clinical suspicion or previous genotyping.
11. Abnormality identified on baseline serology including leukocytosis, leukopenia, thrombocytopenia, anemia, abnormal renal function (Cr > 1.5 x upper limit of normal), or abnormal liver function (ALT, ALP, or AST > 1.5x upper limit of normal)
12. New psychotropic medication (i.e. medication with known or potential impact on psychiatric symptoms, including selective serotonin reuptake inhibitors, benzodiazepines, antipsychotics, stimulants, anticonvulsants, mood stabilizers, or other medications) or other ongoing regular medication started in the 10 weeks prior to baseline, or change in dose in the 4 weeks prior to baseline
13. Changes in CBT or other psychotherapy in the 4 weeks prior to baseline (i.e. change in regular frequency, modality, or care provider)
14. Notable other treatment changes during the study period (either pharmacotherapy or psychotherapy)
15. No regular physician (family doctor or specialist) providing usual medical care
16. Participant/parents unable to provide informed consent or assent or participate in self-care, AE reporting, or follow-up assessments
17. Inability to have blood pressure measured within 2 months prior to enrollment (either on-site at BCCH or by a primary care provider).
18. Intention of pregnancy in participants with child-bearing potential.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Children's Yale-Brown Obsessive-Compulsive Scale, 1st Edition (CY-BOCS-I) | 12 weeks (adjusted for baseline severity)
  The CY-BOCS is a well-validated clinician-rated measure to assess obsessive-compulsive symptom severity. This results in two subscale total scores, Obsessions and Compulsions, each ranging from 0-20, with a higher score indicating greater symptom severity. These subscale scores are summed to provide a total score, ranging from 0 to 40, that is used to measure overall OCD symptom severity.

SECONDARY OUTCOMES:
Children's Yale-Brown Obsessive-Compulsive Scale, 1st Edition (CY-BOCS-I) | 6 weeks (adjusted for baseline severity)
  The CY-BOCS is a well-validated clinician-rated measure to assess obsessive-compulsive symptom severity. This results in two subscale total scores, Obsessions and Compulsions, each ranging from 0-20, with a higher score indicating greater symptom severity. These subscale scores are summed to provide a total score, ranging from 0 to 40, that is used to measure overall OCD symptom severity.
Proportion of participants achieving a clinically meaningful treatment response. | 6 weeks, 12 weeks
  Defined as a 25% reduction in the Children's Yale-Brown Obsessive-Compulsive Scale, 1st Edition (CY-BOCS-I) score or Clinical Global Impression of Improvement (CGI-I) of 1 or 2. As described for the primary outcome measure, this scale has a total score ranging from 0 to 40 with higher scores indicating greater symptom severity.
  The CGI scales includes single item, clinician-rated, Likert-type scales of severity and improvement. The CGI-S (severity) is a frequently-used measure for assessment of symptom severity across multiple psychiatric illnesses due to its face validity and ease of clinical use. Responses range from 1 (no symptoms) through 7 (among the most severely ill patients, extremely severe symptoms, or completely non-functional). The CGI-I (improvement) typically but not always tracks with CGI-S and has been used previously to define response in treatment trials of pediatric OCD. CGI-I scores range from 1 (very much improved) through to 7 (very much worse).
Proportion of participants achieving clinical remission. | 6 weeks, 12 weeks
  Defined based on Children's Yale-Brown Obsessive-Compulsive Scale, 1st Edition (CY-BOCS-I) ≤ 14. As described for the primary outcome measure, this scale has a total score ranging from 0 to 40 with higher scores indicating greater symptom severity.
Mean Clinical Global Impression of Severity (CGI-S) | 6 weeks, 12 weeks (adjusted for baseline)
  As described in Outcome 3, the CGI-S is a 7-point clinician-rated Likert scale with scores ranging from 1 (no OCD symptoms) through 7 (among the most severely ill patients, extremely severe symptoms, or completely non-functional).
Mean Clinician Global Impression of Improvement (CGI-I) | 6 weeks, 12 weeks (adjusted for baseline)
  As described in Outcome 3, the CGI-I is a 7-point clinician-rated Likert scale with scores ranging from 1 (very much improved) through to 7 (very much worse).
Proportion of participants reporting adverse events that are possibly, probably, or definitely related to the study intervention. | 0-12 weeks
  Adverse events will be monitored by clinician interview in addition to a questionnaire adapted from the Safety Monitoring Uniform Research Form (SMURF).

CONTACTS AND LOCATIONS:
Overall Officials: S. Evelyn Stewart, MD, Principal Investigator — University of British Columbia; BC Children's Hospital Research Institute; Clara Westwell-Roper, MD, PhD, Study Chair — University of British Columbia; BC Children's Hospital Research Institute
Locations (1):
- BC Children's Hospital Research Institute, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Westwell-Roper C, Best JR, Elbe D, MacFadden M, Baer S, Tucker L, Au A, Naqqash Z, Lin B, Lu C, Stewart SE. Celecoxib versus placebo as an adjunct to treatment-as-usual in children and youth with obsessive-compulsive disorder: protocol for a single-site randomised quadruple-blind phase II study. BMJ Open. 2022 Jan 31;12(1):e054296. doi: 10.1136/bmjopen-2021-054296. PMID 35105633